CLINICAL TRIAL: NCT03584191
Title: Awareness, Care & Treatment In Obesity Management - An International Observation (ACTION-IO)
Brief Title: Awareness, Care & Treatment In Obesity Management - An International Observation
Acronym: ACTION-IO
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-4449; U1111-1209-6406 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Obesity: General population - potential participants will be recruited using various and numerous general population as appropriate in each country.
  Interventions: Other: No treatment given
- Health Care Professionals: Health Care Professionals include primary care physicians and specialists who treat patients with obesity.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Completion of a survey

SUMMARY:
The purpose of this survey is to collect the data on perceptions, behaviours and awareness related to obesity and obesity management for People with Obesity (PwO) and Health Care Professionals (HCP) treating obesity. Data will be collected via online surveys among each of the respondent groups. The surveys are expected to take approximately 25 minutes to complete and will be unique for PwO and HCP. As a cross-sectional study, there will be no treatment of patients.

ELIGIBILITY:
Inclusion Criteria: - PEOPLE WITH OBESITY - Age at least 18 years, both males and females - On-line consent to participate in study - Lives in one of the participating countries: Italy, Spain, United Kingdom (UK), Brazil, Chile, Mexico, Australia, Israel, Saudi Arabia, United Arab Emirates (UAE), Japan, South Korea - Current Body Mass Index (BMI) (based on self-reported height and weight) greater than or equal to 30 kg/sqm in Italy, Spain, UK, Brazil, Chile, Mexico, Australia, Israel, Saudi Arabia, UAE; current BMI greater than or equal to 25 kg/sqm in Japan and South Korea - HEALTH CARE PROFESSIONALS - Physician - Specialty is NOT plastic surgeon, general surgeon, or bariatric surgeon - Practices in one of the participating countries: Italy, Spain, UK, Brazil, Chile, Mexico, Australia, Israel, Saudi Arabia, UAE, Japan, South Korea - In practice at least 2 years - Spends at least 70 percent of time in direct patient care - Has seen at least 100 patients in past month - Has seen at least 10 patients in past month needing weight management defined as: a patient with a BMI greater than or equal to 30 kg/sqm with or without comorbidities. (BMI greater than or equal to 25 kg/sqm in Japan and South Korea) Exclusion Criteria: - PEOPLE WITH OBESITY - Declines to provide income - Previous participation in this study. Participation is defined as having given online consent in this study - Declines to provide race / ethnicity (in applicable countries) - Currently pregnant - Participates in intense fitness or body building programs - Has had significant, unintentional weight loss (due to major injury, illness, etc.) in the past 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with obesity and health care professionals
Sampling Method: Non-Probability Sample
Enrollment: 17287 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Weight loss motivators | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Multiple Item Selection
Proportion of PwO / patients who made serious weight loss effort | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Numeric Response
Response to weight loss discussions | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Single Item Selection
Effective weight loss methods | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Multiple Item Selection
Obesity attitudes | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - End-anchored 5-point Likert agreement scale (from "1", do not agree at all, to "5" completely agree)
Attitudes toward prescription weight loss medication and surgery | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - End-anchored 5-point Likert agreement scale (from "1", do not agree at all, to "5" completely agree)
Weight loss barriers | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - End-anchored 5-point Likert agreement scale(from "1", do not agree at all, to "5" completely agree)
Obesity and weight management | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - End-anchored 5-point Likert agreement scale(from "1", do not agree at all, to "5" completely agree)
Degree to which healthcare and society is meeting needs of people with obesity | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - End-anchored 5-point Likert needs scale(from "1", do not agree at all, to "5" completely agree)

SECONDARY OUTCOMES:
Top factors for improving weight loss outcomes | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Ranking Exercise
Types of weight management goals | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Multiple Item Selection
Most helpful information for patients for weight loss | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Multiple Item Selection
Responsibility for improving health of people with obesity | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Multiple Item Selection
Most helpful support for weight loss | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Multiple Item Selection
Effectiveness of guidelines for treating obesity | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Fully-anchored 5-point Likert scale (from "1", do not agree at all, to "5" completely agree)
Ways you receive information on weight loss management | Start of interviews day 1 until end of data collection day 90
  Online questionnaire - Multiple Item Selection

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (9):
- Novo Nordisk Investigational Site, Baulkham Hills, New South Wales, Australia
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Polanco, Mexico
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Dubai, United Arab Emirates
- Novo Nordisk Investigational Site, Gatwick, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Caterson ID, Alfadda AA, Auerbach P, Coutinho W, Cuevas A, Dicker D, Hughes C, Iwabu M, Kang JH, Nawar R, Reynoso R, Rhee N, Rigas G, Salvador J, Sbraccia P, Vazquez-Velazquez V, Halford JCG. Gaps to bridge: Misalignment between perception, reality and actions in obesity. Diabetes Obes Metab. 2019 Aug;21(8):1914-1924. doi: 10.1111/dom.13752. Epub 2019 May 3. PMID 31032548
- [Derived] Hughes CA, Ahern AL, Kasetty H, McGowan BM, Parretti HM, Vincent A, Halford JCG. Changing the narrative around obesity in the UK: a survey of people with obesity and healthcare professionals from the ACTION-IO study. BMJ Open. 2021 Jun 30;11(6):e045616. doi: 10.1136/bmjopen-2020-045616. PMID 34193488
- [Derived] Dicker D, Alfadda AA, Coutinho W, Cuevas A, Halford JCG, Hughes CA, Iwabu M, Kang JH, Nawar R, Reynoso R, Rhee N, Rigas G, Salvador J, Sbraccia P, Vazquez-Velazquez V, Caterson ID. Patient motivation to lose weight: Importance of healthcare professional support, goals and self-efficacy. Eur J Intern Med. 2021 Sep;91:10-16. doi: 10.1016/j.ejim.2021.01.019. Epub 2021 Feb 6. PMID 33558163
- [Derived] Alfadda AA, Caterson ID, Coutinho W, Cuevas A, Dicker D, Halford JCG, Hughes CA, Iwabu M, Kang JH, Nawar R, Reynoso R, Rhee N, Rigas G, Salvador J, Vazquez-Velazquez V, Sbraccia P. The 3Ds - Discussion, diagnosis and direction: Elements for effective obesity care by healthcare professionals. Eur J Intern Med. 2021 Sep;91:17-25. doi: 10.1016/j.ejim.2021.01.012. Epub 2021 Jan 23. PMID 33495083
- [Derived] Vazquez-Velazquez V, Laviada-Molina H, Garcia-Garcia E, Sandoval-Diez E, Mancillas-Adame L. Perceptions, Attitudes, and Barriers to Obesity Care in Mexico: Data From the ACTION-IO Study. Obesity (Silver Spring). 2021 Feb;29(2):317-326. doi: 10.1002/oby.23077. PMID 33491317
- [Derived] Dicker D, Kornboim B, Bachrach R, Shehadeh N, Potesman-Yona S, Segal-Lieberman G. ACTION-IO as a platform to understand differences in perceptions, attitudes, and behaviors of people with obesity and physicians across countries - the Israeli experience. Isr J Health Policy Res. 2020 Oct 21;9(1):56. doi: 10.1186/s13584-020-00404-2. PMID 33087177
- [Derived] Sbraccia P, Busetto L, Santini F, Mancuso M, Nicoziani P, Nicolucci A. Misperceptions and barriers to obesity management: Italian data from the ACTION-IO study. Eat Weight Disord. 2021 Apr;26(3):817-828. doi: 10.1007/s40519-020-00907-6. Epub 2020 May 8. PMID 32385580